CLINICAL TRIAL: NCT02737007
Title: A Microdose Study to Describe the Intravenous Pharmacokinetics of GSK3191607 in Healthy Male Subjects Following Administration of [14C]-GSK3191607
Brief Title: A Microdose Study in Healthy Subjects to Describe Intravenous Pharmacokinetics of GSK3191607
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204853
Record Dates: First submitted 2016-03-31; First posted 2016-04-13 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Malaria, Falciparum
Keywords: Malaria; Microdose; GSK3191607
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-GSK3191607 IV Microdose (Experimental): Subjects will receive a single microdose of 100 micrograms (mcg) of [14C]-GSK3191607 by intravenous infusion over 15 minutes on Day 1 of the study.
  Interventions: Drug: [14C]-GSK3191607

INTERVENTIONS:
Drug: [14C]-GSK3191607 — [14C]-GSK3191607 is a solution to be administered intravenously as a single dose infusion over 15 minutes. It is a radio-labeled product; 100 mcg of [14C]-GSK3191607 contains approximately 7.4 kilobecquerel (kBq) of [14C] radioactivity.

SUMMARY:
This is an open-label, single-centre, non-randomized study to investigate the pharmacokinetics of GSK3191607, administered as a single intravenous (IV) dose in healthy male subjects.

Six subjects will be administered an IV microdose of radio-labeled [14C]-GSK3191607. The study will provide an early readout on human pharmacokinetic parameters. The results of this study will be used to estimate the potential duration of anti-parasite effect in humans, define predicted clinical oral doses, and hence inform about the compound's potential safety margin.

Each subject will participate in the study for up to 8 weeks, and will have a screening visit, one treatment period, eight outpatient visits, and a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kg and body mass index (BMI) within the range 19.0-31.0 kilograms per meter squared (kg/m^2) (inclusive).
* Male.
* Subjects with female partners of child bearing potential must use a condom from the time of first dose of study medication until follow-up.
* Capable of giving signed informed consent, which includes compliance with pre-defined requirements and restrictions.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5 times upper limit of normal (ULN) (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Mean QT duration corrected for heart rate by Fridericia's formula (QTcF) > 450 milliseconds (msec).
* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or 12-lead electrocardiogram (ECG).
* At screening, a mean supine blood pressure (BP) that is higher (triplicate measurements at least 2 minutes apart) than 140/90 millimeters of mercury (mmHg).
* At screening, a supine mean pulse rate outside the range 40-90 beats per minute (BPM).
* Subject is mentally or legally incapacitated.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study medication, unless in the opinion of the investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Smoking or use of tobacco products. Urinary cotinine levels indicative of use of tobacco products or nicotine-containing products.
* History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >21 units. One unit is equivalent to 8 grams (g) of alcohol: a half pint (~240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medication or its components, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates the subject's participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months before first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for Human immunodeficiency virus (HIV).
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months before dosing. A subject's previous effective dose will be reviewed by the medical investigator to ensure there is no risk of contamination/carryover into the current study.
* Subjects who have received a total body radiation dose of greater than 5.0 millisieverts (mSv) (upper limit of World Health Organization [WHO] category II) or exposure to significant radiation (for example, serial x ray or Computed Tomography (CT) scans, barium meal, etc.) in the 12 months before dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days before the first dose of study medication until the last study visit.
* The subject has participated in a clinical trial and has received an investigational product within the following time period before the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months before the first dosing day.
* An occupation which requires monitoring for radiation exposure, nuclear medicine procedures or excessive x-rays within the past 12 months before dosing.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of GSK3191607 in plasma following a single intravenous (IV) microdose | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
Terminal phase half life (t1/2) of GSK3191607 following a single IV microdose | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
Time of occurrence of Cmax (tmax) of GSK3191607 following a single IV microdose | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
AUC(0-t) of GSK3191607 following a single IV microdose | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  AUC(0-t) is the area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration.
AUC(0-infinity) of GSK3191607 following a single IV microdose | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  AUC(0-infinity) is the area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time.
Systemic clearance (CL) of GSK3191607 following a single IV microdose | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
GSK3191607 volume of distribution at steady state (Vss) | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
Cmax of radioactive drug-related material (RDM) in plasma following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  RDM is a measure of total radioactivity. Cmax of RDM will be compared with that of the parent drug (GSK3191607).
T1/2 of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  T1/2 of RDM will be compared with that of the parent drug.
Tmax of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  Tmax of RDM will be compared with that of the parent drug.
AUC(0-t) of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  AUC(0-t) of RDM will be compared with that of the parent drug.
AUC(0-infinity) of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  AUC(0-infinity) of RDM will be compared with that of the parent drug.
Amount of RDM excreted in urine (Ae) following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0-24 hours and 24-48 hours after the start of infusion
  Subjects will be asked to void their bladders before study treatment administration. A blank urine sample will be collected pre-dose.

SECONDARY OUTCOMES:
Whole-Blood:Plasma ratio of Cmax of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  Cmax of RDM in whole blood will be compared with that of RDM in plasma.
Whole-Blood:Plasma ratio of tmax of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  Tmax of RDM in whole blood will be compared with that of RDM in plasma.
Whole-Blood:Plasma ratio of t1/2 of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  T1/2 of RDM in whole blood will be compared with that of RDM in plasma.
Whole-Blood:Plasma ratio of AUC(0-t) of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  AUC(0-t) of RDM in whole blood will be compared with that of RDM in plasma.
Whole-Blood:Plasma ratio of AUC(0-infinity) of RDM following a single IV microdose of [14C]-GSK3191607 | Pre-dose; and 0.25, 0.75, 1.5, 3, 6, 8, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, and 336 hours following start of infusion
  AUC(0-infinity) of RDM in whole blood will be compared with that of RDM in plasma.
Number of subjects with adverse events | Start of infusion until follow-up (up to Day 25)
Number of subjects with clinically significant abnormal laboratory parameters | Day -1, Day 1, Day 2, and follow-up (up to Day 25)
  Hematology, clinical chemistry, and urinalysis parameters will be evaluated.
Number of subjects with clinically significant abnormal 12-lead electrocardiogram (ECG) parameters | Pre-dose, Day 1, Day 2, and follow-up (up to Day 25)
  12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Bazett's formula (QTcB) intervals.
Number of subjects with clinically significant abnormal vital signs parameters | Pre-dose, Day 1, Day 2, Day 3, and follow-up (up to Day 25)
  Vital signs will be measured in a semi-supine position after 5 minutes rest and will include systolic and diastolic blood pressure and pulse rate.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 204853 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/204853?search=study&b'search_terms=204853'#rs